CLINICAL TRIAL: NCT04639401
Title: Effect of Motor Entrainment to Auditory Cues and Music During Walking on Quality of Movement and Percieved Fatigue in Persons With Multiple Sclerosis With Cerebellar Lesions
Brief Title: Auditory-motor Coupling in Multiple Sclerosis With Cerebellar Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: National MS Center Melsbroek (Other); Revalidatie & MS Centrum Overpelt (Other)
Responsible Party: Principal Investigator, Peter Feys, Principal Investigator, Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AMCiMS-001
Record Dates: First submitted 2020-11-09; First posted 2020-11-20 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis; Cerebral Lesion
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- persons with Multiple Sclerosis (Experimental)
  Interventions: Other: motor entrainment to auditory cues and music during walking on quality of movement
- Healthy controls (Placebo Comparator)
  Interventions: Other: motor entrainment to auditory cues and music during walking on quality of movement

INTERVENTIONS:
Other: motor entrainment to auditory cues and music during walking on quality of movement — The study contains 1 descriptive and 4 experimental sessions. In the descriptive session, participant's clinical motor and cognitive functions are collected. In the first experimental session, participant's beat perception and synchronisation abilities is examined within a finger tapping paradigm. In the following experimental sessions participants synchronsiation abilities is examined during walking paradigms, to music and metronomes, at different tempi and alignment strategies. In the latter three sessions, apart from outcome measures of synchronization the following will be collected as well: spatio-temporal gait parameters, perceived fatigue, perceived motivation and perceived speed of walking.

SUMMARY:
This study is a case-control observational study, involving persons with multiple sclerosis and healthy controls. The study contains 1 descriptive and 4 experimental sessions. In the descriptive session, participant's clinical motor and cognitive functions are collected. In the first experimental session, participant's beat perception and synchronisation abilities is examined within a finger tapping paradigm. In the following experimental sessions participants synchronsiation abilities is examined during walking paradigms, to music and metronomes, at different tempi and alignment strategies. In the latter three sessions, apart from outcome measures of synchronization the following will be collected as well: spatio-temporal gait parameters, perceived fatigue, perceived motivation and perceived speed of walking.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Multiple sclerosis >1 year,
* type of lesions: cerebellar lesions,
* walking speed 0.8-1.2m/s, ability to walk for 6 minutes continuously (canes and rollators are permitted).

Exclusion Criteria:

* relapse 3 months prior to enrollment,
* cognitive impairment impeding understanding of instructions,
* beat amusia,
* deafness,
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Resultant Vector Length | week 3
  synchronisation consistency
Resultant Vector Length | week 4
  synchronisation consistency
Resultant Vector Length | week 5
  synchronisation consistency
Relative phase angle | week 3
  asynchrony in time to quantify synchronization accuracy (in degrees and in milliseconds respectively)
Relative phase angle | week 4
  asynchrony in time to quantify synchronization accuracy (in degrees and in milliseconds respectively)
Relative phase angle | week 5
  asynchrony in time to quantify synchronization accuracy (in degrees and in milliseconds respectively)
Perceptual tempo and rhythm judgements | week 2
  subjective indications in regards to what the participants hear in terms
Asynchrony | week2
  timing difference between the tap and the beat
EEG | week 2
  64 channel EEG measurement (only conducted in 4 PwMS and HC) -> neural correlates of entrainment
Muscle weakness | week 1
  Motricity Index of dorsi flexors, knee extensors and hip flexors -
Spasticity | week 1
  Modified Aschowrth scale Hamstrings, Tricepts Surae, Quadricepts
Ataxia | week 1
  Scale for the assessment and rating of ataxia
Dynamic gait index | week 1
  dynamic balance
Time up and Go test | week 1
  balance
6 minute walking test | week 1
  gait pattern and endurance
Brief repeatable battery of Rao | week 1
  cognitive test
Symbol digit mobility test | week 1
  cognitive test
Stroop test 0 | week 1
  cognitive test
MS walking scale -12 | week 1
  impact of MS on walking ability
Activities-specific balance confidence scale | week 1
  rating of balance confidence in performing activities of daily life
Modified fatigue impact scale | week 1
  effect of fatigue
Hospital Anxiety and Depression Scale | week 1
  determine the levels of anxiety and depression
Dual task questionnaire | week 1
  troubles a person have when performing a dual task during daily activity

SECONDARY OUTCOMES:
Cadence | week 3
  number of steps per minute
Cadence | week 4
  number of steps per minute
Cadence | week 5
  number of steps per minute
Stride length | week 3
  distance between consecutive steps (cm)
Stride length | week 4
  distance between consecutive steps (cm)
Stride length | week 5
  distance between consecutive steps (cm)
speed | week 3
  gait velocity (m/s)
speed | week 4
  gait velocity (m/s)
speed | week 5
  gait velocity (m/s)
Double Support | week 3
  time that both legs are in contact with the floor (mseconds)
Double Support | week 4
  time that both legs are in contact with the floor (mseconds)
Double Support | week 5
  time that both legs are in contact with the floor (mseconds)
Perceived cognitive and physical fatigue | week 3
  A visual analogue scale will be used, and participants will be asked to rate their perceived cognitive and physical fatigue levels before and after each experimental walking conditions
Perceived cognitive and physical fatigue | week 4
  A visual analogue scale will be used, and participants will be asked to rate their perceived cognitive and physical fatigue levels before and after each experimental walking conditions
Perceived cognitive and physical fatigue | week 5
  A visual analogue scale will be used, and participants will be asked to rate their perceived cognitive and physical fatigue levels before and after each experimental walking conditions
Perceived motivation | week 3
  A Likert scale will be used, and participants will be asked to rate their perceived motivation of walking after each experimental walking conditions
Perceived motivation | week 4
  A Likert scale will be used, and participants will be asked to rate their perceived motivation of walking after each experimental walking conditions
Perceived motivation | week 5
  A Likert scale will be used, and participants will be asked to rate their perceived motivation of walking after each experimental walking conditions
Perceived walking speed | week 3
  A Likert scale will be used, and participants will be asked to rate their perceived walking speed relative to their usual walking after each experimental walking conditions
Perceived walking speed | week 4
  A Likert scale will be used, and participants will be asked to rate their perceived walking speed relative to their usual walking after each experimental walking conditions
Perceived walking speed | week 5
  A Likert scale will be used, and participants will be asked to rate their perceived walking speed relative to their usual walking after each experimental walking conditions

CONTACTS AND LOCATIONS:
Overall Officials: Peter Feys, prof. dr., Principal Investigator — Hasselt University; Lousin Moumdjian, dr., Study Chair — Hasselt University
Locations (2):
- Belgium (2):
  - National MS Center Melsbroek, Melsbroek
  - Noorderhart Revalidatie & MS centrum, Overpelt

IPD SHARING:
Plan to Share IPD: No